CLINICAL TRIAL: NCT01198249
Title: A Randomized, Open Label, Multiple Dose, Crossover Study to Investigate Pharmacokinetic Drug Interactions Between Single and Concomitant Administrations of Amlodipine, Losartan, and Hydrochlorothiazide(HCTZ) in Subjects With (Pre)Hypertension
Brief Title: Pharmacokinetic Drug Interactions Between Single and Concomitant Administrations of Amlodipine, Losartan, and Hydrochlorothiazide in Subjects With (Pre)Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Kyung-Mi Park / Director, Hanmi Pharmaceutial Co., Ltd.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 4-2010-0295
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Losartan; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- amlodipine monotherapy (Experimental)
  Interventions: Drug: multiple dose, crossover study between single and concomitant administrations of amlodipine, losartan, and hydrochlorothiazide
- losartan monotherapy (Experimental)
  Interventions: Drug: multiple dose, crossover study between single and concomitant administrations of amlodipine, losartan, and hydrochlorothiazide
- HCTZ (Experimental)
  Interventions: Drug: multiple dose, crossover study between single and concomitant administrations of amlodipine, losartan, and hydrochlorothiazide
- mlodipine and Losartan and HCTZ (Experimental)
  Interventions: Drug: multiple dose, crossover study between single and concomitant administrations of amlodipine, losartan, and hydrochlorothiazide

INTERVENTIONS:
Drug: multiple dose, crossover study between single and concomitant administrations of amlodipine, losartan, and hydrochlorothiazide — amlodipine 10 mg for 9 days , losartan 100 mg for 9 days, hydrochlorothiazide (HCTZ) 25 mg for 9 days and combination of amlodipine 10 mg, losartan 100 mg and hydrochlorothiazide (HCTZ) 25 mg for 9 days, 4 way crossover study

SUMMARY:
This study is aimed to evaluate the pharmacokinetics and the drug-drug interaction among anti-hypertension drugs-amlodipine, losartan, and hydrochlorothiazide. This pilot study provides useful information to develop a new fixed dose combination drug.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects 20-50 years of age
* Above 55Kg and within ±20% ideal body weight
* Subjects who are in average of 130mmHg ≤ systolic blood pressure (SBP) < 160mmHg, 80mmHg ≤ diastolic blood pressure (DBP) < 100mmHg
* Female subject who confirmed non-pregnant status and agree to comply with proper contraception.
* Subjects who wrote informed consent

Exclusion Criteria:

* Subjects who are suspected to have acute disease
* Subjects who have past history that may affect drug absorption, distribution, metabolism and elimination
* Subjects who have gastrointestinal history
* Subjects whose heartrate is less than 60
* Subject who suspected to orthostatic hypotension
* Subjects who have clinically significant allergy disease
* Subject is currently participating or has participating in a study with an investigational compound or device within 30 days of signing informed consent
* Administration of prescription drug within 14 days or over the counter (OTC) drug within 7 days
* Subjects who have past history of drug abuse and positive in drug screening test
* Subjects who donate whole blood within 60 days and platelet within 30days.
* Subjects taking St John's wort or CYP inhibitor and inducer

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2010-09; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Yong Chung, MD, Ph.D, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea